CLINICAL TRIAL: NCT01386606
Title: A Randomized, Single Blind, Multi-Center Phase II Study to Evaluate the Effect of Three Different Doses of Androxal and AndroGel on 24-Hour Luteinizing Hormone and Testosterone in Normal Healthy Men
Brief Title: The Effect on Androxal Versus Androgel on Morning Testosterone in Men With Secondary Hypogonadism (Low Testosterone)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZA-204
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Results first posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-08

CONDITIONS: Secondary Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene; Testosterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Androxal 6.25 mg (Experimental): Androxal 6.25 mg/day
  Interventions: Drug: Androxal (enclomiphene citrate)
- Androxal 12.5 mg (Experimental): Androxal 12.5 mg/day
  Interventions: Drug: Androxal (enclomiphene citrate)
- Androxal 25 mg (Experimental): Androxal 25 mg/day
  Interventions: Drug: Androxal (enclomiphene citrate)
- AndroGel (Active Comparator): AndroGel 5G topical testosterone
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Androxal (enclomiphene citrate) — capsule oral
  1X a day 6 weeks
  Other Names: Androxal; low testosterone therapy
  Arms: Androxal 12.5 mg; Androxal 25 mg; Androxal 6.25 mg
Drug: Testosterone — topical gel
  1X a day 6 weeks
  Other Names: topical testosterone; testosterone gel; exogenous testosterone
  Arms: AndroGel

SUMMARY:
The study will determine the effects of three doses of Androxal(enclomiphene citrate)on morning testosterone versus AndroGel(approved topical treatment)in men with low testosterone (<350 ng/dL)after 6 weeks of continuous dosing.

DETAILED DESCRIPTION:
Study will require 7 visits, which includes 2 overnight stays in a clinic. One visit is an eye exam. Blood samples are required at all visits including sampling every hour for a 24 hour time period during the 2 overnight stays. A six month extension study will be available for all subjects completing the 6-week study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between the ages of 18 and 65 years of age exhibiting morning testosterone ≤350 ng/dL.
* All clinical laboratory tests within normal ranges (any clinically significant deviation of laboratory results will require approval of sponsor)
* Ability to complete the study in compliance with the protocol
* Ability to understand and provide written informed consent
* Agreement to use a condom, and with a fertile female partner, another form of contraception.
* Agreement to provide a semen sample in the clinic

Exclusion Criteria:

* Use of an injectable, oral, topical, or subcutaneous pelleted testosterone within 3 months prior to study
* Use of spironolactone, cimetidine, 5α-reductase inhibitors, hCG, androgen, estrogen, anabolic steroid, DHEA, or herbal hormone products during the study
* Use of Clomid in the past year or during the study
* Uncontrolled hypertension or diabetes mellitus based on the Investigator's assessment at baseline. Subjects treated for Type II diabetes but exhibiting glycemic control will be allowed into the study. Newly diagnosed diabetics need to be treated for at least 48 hours before being enrolled in the study.
* A hematocrit ≥51 % or a hemoglobin ≥17 g/dL
* Clinically significant abnormal findings on screening examination
* Use of an investigational drug or product, or participation in a drug or medical device research study within 30 days prior to receiving study medication
* Known hypersensitivity to Clomid
* Any condition which in the opinion of the investigator would interfere with the participant's ability to provide informed consent, comply with study instructions, possibly confound interpretation of study results, or endanger the participant if he took part in the study
* Irreversibly infertile or compromised fertility (cryptorchism, Kallman Syndrome, primary hypogonadism, vasectomy, or tumors of the pituitary)
* History of breast cancer
* History of prostate cancer or a suspicion of prostate disease unless ruled out by prostate biopsy, or a PSA >3.6
* History of known hyperprolactinemia with or without a tumor
* Chronic use of medications use such as glucocorticoids
* Chronic use of narcotics
* Subjects known to be positive for HIV
* Subjects with end stage renal disease
* Subjects with cystic fibrosis (mutation of the CFTR gene)
* Subjects unable to provide a semen sample in the clinic
* Subject has a BMI >42 kg/m2

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jolene Berg, MD, Principal Investigator — Cetero Research, San Antonio
Locations (2):
- United States (2):
  - Centex Research, Houston, Texas
  - Cetero Research, San Antonio, Texas

REFERENCES:
- See also: Sponsor website — http://www.reprosrx.com
- See also: Related Info — http://www.helpmylowT.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Androxal 6.25 mg; Androxal 12.5 mg; Androxal 25 mg: enclomiphene citrate: capsule oral
  1X a day 6 weeks
- AndroGel: AndroGel 5G topical testosterone
  Testosterone: topical gel
  1X a day 6 weeks
Period: Overall Study
Arm/Group | Androxal 6.25 mg | Androxal 12.5 mg | Androxal 25 mg | AndroGel
Started | 16 | 14 | 16 | 14
Completed | 12 | 10 | 13 | 13
Not Completed | 4 | 4 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Subject incarcerated | 0 | 1 | 0 | 0
Not completed — Unable to draw PK | 1 | 0 | 0 | 0
Not completed — T levels too high | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis consisted of all subjects enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Androxal 6.25 mg | Androxal 12.5 mg | Androxal 25 mg | AndroGel | Total
Number analyzed (Participants) | 16 | 14 | 16 | 14 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (8.8) | 51.7 (9.2) | 51.8 (13.0) | 53.5 (9.8) | 52.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 16 | 14 | 16 | 14 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 8 | 10 | 2 | 28
  White | 8 | 6 | 6 | 12 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 16 | 14 | 60
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 33.3 (5.9) | 31.2 (6.6) | 31.6 (6.3) | 31.0 (6.1) | 31.8 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Average and Maximum Testosterone Concentration
Description: The primary efficacy endpoint will be 24-hour average (TTavg) and maximum (TTmax) testosterone concentration compared to baseline after 6 weeks of treatment.
  Time points (in hours after dosing) at which testosterone concentration was measured are: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24.
Time Frame: Baseline and Week 6
Population: ITT, subjects who received at least one dose of study drug and had at least one post-dose efficacy measure.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Androxal 6.25 mg | Androxal 12.5 mg | Androxal 25 mg | AndroGel
Number analyzed (Participants) | 12 | 10 | 13 | 13
ng/dL
  TTavg at Baseline | 262.3 (80.3) | 373.6 (172.1) | 298.3 (100.5) | 322.4 (102.9)
  TTavg at Week 6 | 392.4 (152.6) | 460.8 (129.1) | 586.7 (142.4) | 543.9 (229.8)
  TTmax at Baseline | 358.5 (120.5) | 513.7 (222.2) | 425.9 (114.3) | 562.3 (488.5)
  TTmax at Week 6 | 524.5 (178.7) | 607.5 (167.7) | 764.3 (158.7) | 930.1 (550.4)
Statistical Analysis 1: Comparison: Androxal 6.25 mg vs Androxal 12.5 mg vs Androxal 25 mg vs AndroGel; Regression of 24 Hours Average Total Testosterone, Treatment Group and Morning Testosterone at Week 6. Modeling 24 hour average total testosterone by morning testosterone and treatment group; Test type: Superiority or Other; p = 0.056, Regression, Linear — P-value of treatment group
Statistical Analysis 2: Comparison: Androxal 6.25 mg vs Androxal 12.5 mg vs Androxal 25 mg vs AndroGel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.436, Regression, Linear — P-value for Androxal 25 mg treatment group; Regression Coefficient = -45.77, 95% CI 2-sided [-143.5 to 51.98]
Statistical Analysis 3: Comparison: Androxal 6.25 mg vs Androxal 12.5 mg vs Androxal 25 mg vs AndroGel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.068, Regression, Linear — P-value for Androxal 12.5 mg group; Regression Coefficient = -110.9, 95% CI 2-sided [-210.6 to -11.23]
Statistical Analysis 4: Comparison: Androxal 6.25 mg vs Androxal 12.5 mg vs Androxal 25 mg vs AndroGel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.011, Regression, Linear — P-value for Androxal 6.25 mg group; Regression Coefficient = -148.5, 95% CI 2-sided [-242.9 to -54.05]
Statistical Analysis 5: Comparison: Androxal 6.25 mg vs Androxal 12.5 mg vs Androxal 25 mg vs AndroGel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Linear — P-value for morning total testosterone (adjusted for treatment effect if treatment group is significant); Regression Coefficient = 0.58, 95% CI 2-sided [0.37 to 0.79]

2. Secondary Outcome: Change in Leuteinizing Hormone (LH)
Description: Changes in morning LH after continuous dosing
Time Frame: Baseline, Week 2, Week 4, Week 6
Population: ITT, subjects who received at least one dose of study drug and had at least one post-dose efficacy measure.
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Androxal 6.25 mg | Androxal 12.5 mg | Androxal 25 mg | AndroGel
Number analyzed (Participants) | 15 | 13 | 16 | 14
mIU/mL
  Morning LH at Baseline | 3.63 (1.55) | 4.82 (1.63) | 4.98 (3.45) | 3.57 (2.23)
  Morning LH at Week 2 | 5.49 (2.69) | 8.60 (4.11) | 9.64 (5.04) | 2.00 (2.12)
  Morning LH Change from Baseline at Week 2 | 1.99 (2.38) | 3.78 (3.29) | 4.66 (3.56) | -1.57 (2.20)
  Morning LH at Week 4 | 6.92 (3.59) | 7.20 (2.97) | 11.78 (7.39) | 1.88 (2.68)
  Morning LH Change from Baseline at Week 4 | 3.43 (3.20) | 2.38 (3.54) | 6.79 (5.54) | -1.69 (1.58)
  Morning LH at Week 6 | 6.1 (3.3) | 8.2 (3.3) | 14.5 (10.5) | 2.2 (2.8)
  Morning LH Change from Baseline at Week 6 | 2.60 (3.32) | 3.39 (3.37) | 9.51 (8.15) | -1.41 (2.01)
Statistical Analysis 1: Comparison: Androxal 6.25 mg vs Androxal 12.5 mg vs Androxal 25 mg vs AndroGel; ANOVA results - change from baseline in morning LH at Week 2. Modeling change from baseline by treatment group; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for treatment group effect
Statistical Analysis 2: Comparison: Androxal 6.25 mg vs Androxal 12.5 mg vs Androxal 25 mg vs AndroGel; ANOVA results - change from baseline in morning LH at Week 4. Modeling change from baseline by treatment group; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for treatment group effect
Statistical Analysis 3: Comparison: Androxal 6.25 mg vs Androxal 12.5 mg vs Androxal 25 mg vs AndroGel; ANOVA results - change from baseline in morning LH at Week 6. Modeling change from baseline by treatment group; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for treatment group effect

3. Post Hoc Outcome: Morning Testosterone Correlated With Serial Testosterone.
Description: 9 AM morning testosterone correlated with Week 6 serial testosterone Cavg, Cmin, and Cmax.
  If a subject did not have a Week 6 serial testosterone Cavg, Cmin, or Cmax then they were not included for that particular correlation calculation.
Time Frame: Week 6
Population: All Androxal subjects with Week 6 serial testosterone measurements.
Measure: Number; unit: Number of Subjects
Groups:
- Androxal Pooled Dose Levels: Androxal 6.25, 12.5, and 25 mg subjects combined into a single group.
Arm/Group | Androxal Pooled Dose Levels
Number analyzed (Participants) | 35
Number of Subjects | 35
Statistical Analysis 1: Comparison: Androxal Pooled Dose Levels; Pearson correlation between 9 am morning testosterone and serial testosterone Cavg at Week 6; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Pearson Correlation = 0.90993
Statistical Analysis 2: Comparison: Androxal Pooled Dose Levels; Pearson correlation between 9 am morning testosterone and serial testosterone Cmin at Week 6; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Pearson Correlation = 0.86541
Statistical Analysis 3: Comparison: Androxal Pooled Dose Levels; Pearson correlation between 9 am morning testosterone and serial testosterone Cmax at Week 6; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Pearson Correlation = 0.89643

4. Other Pre Specified Outcome: Enclomiphene Pharmacokinetic Parameters at Week 6 - Cmax.
Description: The Cmax for plasma concentration.
Time Frame: Week 6
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Androxal 6.25 mg: Androxal 6.25 mg/day
  Androxal (enclomiphene citrate): capsule oral
  1X a day 6 weeks
- Androxal 12.5 mg: Androxal 12.5 mg/day
  Androxal (enclomiphene citrate): capsule oral
  1X a day 6 weeks
- Androxal 25 mg: Androxal 25 mg/day
  Androxal (enclomiphene citrate): capsule oral
  1X a day 6 weeks
Arm/Group | Androxal 6.25 mg | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 12 | 10 | 13
ng/mL | 1.8154 (0.8358) | 3.3899 (2.0239) | 16.2993 (12.8952)

5. Secondary Outcome: Change in Follicle Stimulating Hormone (FSH)
Description: Changes in morning FSH after continuous dosing
Time Frame: Baseline, Week 2, Week 4, Week 6
Population: ITT, subjects who received at least one dose of study drug and had at least one post-dose efficacy measure.
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Androxal 6.25 mg | Androxal 12.5 mg | Androxal 25 mg | AndroGel
Number analyzed (Participants) | 15 | 13 | 16 | 14
mIU/mL
  Morning FSH at Baseline | 4.61 (1.97) | 5.63 (2.26) | 6.31 (4.28) | 6.38 (2.79)
  Morning FSH at Week 2 | 6.18 (2.56) | 7.77 (3.03) | 11.41 (8.19) | 3.80 (3.06)
  Morning FSH Change from Baseline at Week 2 | 1.60 (1.73) | 2.14 (2.15) | 5.09 (4.32) | -2.58 (1.84)
  Morning FSH at Week 4 | 6.45 (2.70) | 7.12 (2.66) | 12.34 (9.59) | 3.72 (3.66)
  Morning FSH Change from Baseline at Week 4 | 1.66 (1.94) | 1.48 (2.58) | 6.03 (5.90) | -2.66 (2.20)
  Morning FSH at Week 6 | 5.69 (3.34) | 8.19 (3.25) | 13.45 (10.84) | 3.35 (3.34)
  Morning FSH Change from Baseline at Week 6 | 1.42 (2.53) | 2.56 (2.53) | 7.14 (7.19) | -3.03 (2.21)
Statistical Analysis 1: Comparison: Androxal 6.25 mg vs Androxal 12.5 mg vs Androxal 25 mg vs AndroGel; ANOVA results - change from baseline in morning FSH at Week 2. Modeling change from baseline by treatment group; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for treatment group effect
Statistical Analysis 2: Comparison: Androxal 6.25 mg vs Androxal 12.5 mg vs Androxal 25 mg vs AndroGel; ANOVA results - change from baseline in morning FSH at Week 4. Modeling change from baseline by treatment group; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for treatment group effect
Statistical Analysis 3: Comparison: Androxal 6.25 mg vs Androxal 12.5 mg vs Androxal 25 mg vs AndroGel; ANOVA results - change from baseline in morning FSH at Week 6. Modeling change from baseline by treatment group; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for treatment group effect

6. Other Pre Specified Outcome: Enclomiphene Pharmacokinetic Parameters at Week 6 - Tmax.
Description: The Tmax for plasma concentration.
Time Frame: Week 6
Population: PK population
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Androxal 6.25 mg | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 12 | 10 | 13
h | 2.33 (0.98) | 2.42 (1.21) | 2.41 (1.48)

7. Other Pre Specified Outcome: Enclomiphene Pharmacokinetic Parameters at Week 6 - AUC0-24.
Description: The area under the curve for plasma concentration over time from zero to 24 hours (AUC0-24).
Time Frame: Week 6
Population: PK population
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Androxal 6.25 mg | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 12 | 10 | 13
ng*h/mL | 21.200 (14.399) | 34.012 (21.419) | 150.51 (132.32)

ADVERSE EVENTS:
Arm/Group | Androxal 6.25 mg | Androxal 12.5 mg | Androxal 25 mg | AndroGel
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 2/16 | 1/14 | 1/16 | 4/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Androxal 6.25 mg (N=16) | Androxal 12.5 mg (N=14) | Androxal 25 mg (N=16) | AndroGel (N=14)
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Defaecation urgency (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Irritability (General disorders) | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Allodynia (Nervous system disorders) | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Libido increased (Psychiatric disorders) | 0 | 0 | 0 | 1
Urinary hesitancy (Renal and urinary disorders) | 0 | 1 | 0 | 0
Epididymal cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights.